CLINICAL TRIAL: NCT03217578
Title: Study on the Neonatal Screening of Spinal Muscular Atrophy
Brief Title: Neonatal Spinal Muscular Atrophy (SMA) Screening
Acronym: SMA
Status: Recruiting | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: The Chinese Foundation of Health (Unknown); Taipei Institute of Pathology (Other Government)
Responsible Party: Sponsor
Other Study IDs: SMA-NBS001
Record Dates: First submitted 2017-07-12; First posted 2017-07-14 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-01

CONDITIONS: Spinal Muscular Atrophy
Keywords: Spinal Muscular Atrophy; Newborn Screening
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: SMA Newborn Screening

SUMMARY:
Parents or legal guardian of neonates who signed agreement will receive SMA screening test if their neonates are affected with SMA. The dried blood spots of routine newborn screening samples will be used to test if neonates have lost 2 copies of SMN1 gene. If neonates have positive SMA screening test, further confirmation with multiplex ligation-dependent probe amplification (MLPA) test and prospective motor function monitoring including physical and neurological examinations will be proved to make SMA confirmation. For any confirmed SMA patient, genetic counseling and standard of care will be proved.

ELIGIBILITY:
Inclusion Criteria:

1. Neonates born in Taiwan who receive regular newborn screening suggested by Ministry of Heath and Welfare.
2. Parents or legal guardian agree to perform SMA newborn screening.

Exclusion Criteria:

Parents or legal guardian do not agree to perform SMA newborn screening.

Ages: 0 Weeks to 2 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Neonates whose parents agree to be tested.
Sampling Method: Probability Sample
Enrollment: 250000 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of neonates with confirmed the deletion of 2 copies of SMN1 gene | 3 years
  Neonates with positive SMA newborn screening will be confirmed by multiplex ligation-dependent probe amplification (MLPA) test

SECONDARY OUTCOMES:
Number of neonates with confirmed SMA | 3 years
  Neonates with confirmed the deletion of 2 copies of SMN1 gene by MLPA test will be followed till SMA symptoms appear.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available